CLINICAL TRIAL: NCT00823732
Title: Palliative Care for Quality of Life and Symptom Concerns in Late Stage Lung Cancer
Brief Title: Effects of Palliative Care on Quality of Life and Symptom Control in Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08035; P01CA136396 (NIH); P30CA033572 (NIH); CHNMC-08035; CDR0000631258 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Early Intervention, Educational; Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 2 Intervention (Active Comparator): GROUP II (palliative care intervention): Patients receive an individualized interdisciplinary palliative care intervention comprising learner-centered, knowledge-centered, assessment-centered, and community-centered concepts. Patients undergo 4 teaching sessions, focused on physical, psychological, social, and spiritual well-being, once weekly in weeks 3-6. Patients then receive 4 follow-up phone calls in weeks 9, 13, 17, and 21.
  Interventions: Other: educational intervention; Other: medical chart review; Other: questionnaire administration; Procedure: end-of-life treatment/management; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment; Procedure: management of therapy complications; Procedure: assessment of therapy complications
- Phase I Usual Care (No Intervention): GROUP I (usual care): Patients receive standard care.

INTERVENTIONS:
Other: educational intervention — Undergo individualized interdisciplinary palliative care intervention
  Arms: Phase 2 Intervention
Other: medical chart review — Ancillary studies
  Arms: Phase 2 Intervention
Other: questionnaire administration — Ancillary studies
  Arms: Phase 2 Intervention
Procedure: end-of-life treatment/management — Undergo end-of-life treatment/management
  Arms: Phase 2 Intervention
Procedure: psychosocial assessment and care — Undergo psychosocial assessment and care
  Arms: Phase 2 Intervention
Procedure: quality-of-life assessment — Ancillary studies
  Arms: Phase 2 Intervention
Procedure: management of therapy complications — Undergo management of therapy complications
  Other Names: complications of therapy, management of
  Arms: Phase 2 Intervention
Procedure: assessment of therapy complications — Undergo assessment of therapy complications
  Arms: Phase 2 Intervention

SUMMARY:
RATIONALE: Palliative care may be more effective than standard care in improving quality of life and symptoms in patients with lung cancer.

PURPOSE: This clinical trial is studying the effects of palliative care on quality of life and symptom control in patients with stage IIIB or stage IV non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the effects of palliative care intervention (PCI) vs standard care on overall quality of life and psychological distress in patients with unresectable stage IIIB or IV non-small cell lung cancer.
* To compare symptom control in these patients.
* To compare geriatric assessment outcomes, as measured by OARS Instrumental Activities of Daily Living, MOS Activities of Daily Living, MOS Social Activities Limitation Scale, Hospital Anxiety and Depression Scale scores, and Karnofsky performance scale, in these patients.
* To compare the effects of the PCI vs standard care on resource use.
* To identify subgroups of patients who benefit most from the PCI in relation to sociodemographic characteristics, treatment factors, and geriatric assessment predictors at week 12.

OUTLINE: Patients are assigned to 1 of 2 groups.

Group I (usual care): Patients receive standard care.

Group II (palliative care intervention): Patients receive an individualized interdisciplinary palliative care intervention comprising sessions, focused on physical, psychological, social, and spiritual well-being, once weekly in weeks 3-6. Patients then receive 4 follow-up phone calls in weeks 9, 13, 17, and 21.

ELIGIBILITY:
Criteria:

* Diagnosis of stage IIIb-IV unresectable NSCLC
* Undergoing treatment with chemotherapy, radiation, or combined modalities
* Living within a 50 mile radius of the City of Hope
* No previous cancer within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Overall quality of life and psychological distress | 6 months after study enrollment
Symptom control | 6 months after study enrollment
Geriatric assessment outcomes as measured by OARS Instrumental Activities of Daily Living, MOS Activities of Daily Living, MOS Social Activities Limitation Scale, Hospital Anxiety and Depression Scale scores, and Karnofsky performance scale | 6 months after study enrollment
Resource use as measured by chart audits | 6 months after study enrollment
Identification of subgroups of patients who benefit most from the palliative care intervention in relation to sociodemographic characteristics, treatment factors, and geriatric assessment predictors at week 24 | Week 24 after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States